CLINICAL TRIAL: NCT03516396
Title: Community Development and Nutrition Education in Banke District, Nepal: Effect on Child Health and Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Heifer Project International (Other)
Responsible Party: Principal Investigator, Laurie Miller, MD, Professor of Pediatrics, Tufts University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AID-OAA-L-1-00006
Record Dates: First submitted 2018-04-09; First posted 2018-05-04 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Malnutrition
Keywords: Nepal; child growth; nutrition education; community development
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized cluster design of households in rural Nepal. Groups will be randomized to receive either: (a) Training Only (livestock management and child nutrition), (b) Training plus enhanced community development activities, or (c) no inputs (Control). After 24 months, groups A and C will receive community development inputs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training Plus (Experimental): Intervention: Community Development
  Training plus enhanced community development activities
  Interventions: Behavioral: Training Plus
- Control (Active Comparator): No inputs
  Interventions: Behavioral: No Inputs then Community development and training
- Training Only (Experimental): Intervention: Training
  Training Only (livestock management and child nutrition)
  Interventions: Behavioral: Training Only

INTERVENTIONS:
Behavioral: Training Plus — Training plus enhanced community development activities
  Arms: Training Plus
Behavioral: Training Only — Training Only (livestock management and child nutrition) for 24 months then add community development inputs
  Arms: Training Only
Behavioral: No Inputs then Community development and training — No inputs for 24 months then add community development and training
  Arms: Control

SUMMARY:
Heifer Project International is a globally active NGO with more than 400 projects in over 30 countries. The organization uses the introduction of livestock and related training in the development of social capital as tools for poverty alleviation, citizen empowerment, and community development. In a pilot project conducted in 2009-2012, these activities were found to promote some improvement in child health and nutritional status. However, robust enhancement of these important indicators was not observed. Heifer now intends to investigate the efficacy of a nutrition and child health education program in amplifying these effects.

DETAILED DESCRIPTION:
Child health and survival remain significant challenges in Nepal. Nepal is ranks 63rd highest in the world for "under 5 mortality" rate, with 54/1000 children dying before their 5th birthdays and 46/1000 infants dying before their first birthdays. Annually, more than 47,000 children die before reaching age 5 years. At these mortality levels, one in every 22 Nepalese children dies before reaching age 1, and one in every 19 does not survive to his or her fifth birthday. Nutritional status of children is extremely poor, with ~29% of children underweight and 41% stunted (respectively, weight and height <-2 SD from median) (UNICEF, 2011) (Ministry of Health and Population et al., 2012).

Heifer Project International is a globally active NGO with more than 400 projects in over 30 countries. The organization uses the introduction of livestock and related training in the development of social capital as tools for poverty alleviation, citizen empowerment, and community development. Heifer International recognizes the links between poverty, child malnutrition, and disease. However, improving economic indicators is not always sufficient to improve child outcomes. Thus, the organization now wishes to conduct a systematic assessment to evaluate the effects of introducing a child health and nutrition component into their work, and to clarify the links (if any) between social capital training and child growth and health. In doing so, Heifer International expects to develop a model which could be adapted for use in other regions of the world. The interaction of Heifer community development activities, specific child and family characteristics, and child health and nutritional status will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* child in household in designated study area of Nepal, age 1 month to 12 years
* family agrees to enrollment

Exclusion Criteria:

* parent refuse to enroll child

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in prevalence of child wasting | baseline, and then at each study visit (every 6 months over 36 months)
  measurement of child's weight in kg and height in cm. These measurements will be converted respectively to weight z scores, height z scores and then weight-for-height z scores using World Health Organization standards. The proportion of wasted children (z score <-2) will be determined.

SECONDARY OUTCOMES:
child health | at each study visit (every 6 months over 36 months)
  Mothers will report the frequency that their child experienced respiratory infection, diarrhea, and/or fever within the 2 weeks prior to the study visit. The presence or absence of each of these symptoms will be scored as either "0" or "1", respectively. These totals will be summed to provide a "health score".
household socioeconomic (SES) status | at each study visit (every 6 months over 36 months)
  Household possessions will be enumerated (e.g., the presence or absence of such items as refrigerator, telephone, car, computer, radio, television). Using principal components analysis, a household SES score will be calculated.
child developmental status | at one study visit each year, starting 12 months after randomization, then annually
  Developmental status of children 66 months of age will be ascertained using the Ages and Stages Questionnaire (for ages 24-66 months). This test combines observation and parent report.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie C Miller, MD, Principal Investigator — Tufts University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Miller LC, Neupane S, Joshi N, Lohani M, Rogers BL, Neupane S, Ghosh S, Webb P. Multisectoral community development in Nepal has greater effects on child growth and diet than nutrition education alone. Public Health Nutr. 2020 Jan;23(1):146-161. doi: 10.1017/S136898001900260X. Epub 2019 Sep 23. PMID 31544735

DOCUMENTS (2):
  • Study Protocol (2014-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03516396/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03516396/SAP_001.pdf